CLINICAL TRIAL: NCT07352683
Title: TAP-blockad Vid öppen Bukkirurgi Hos Barn
Brief Title: Open TAP-block in Pediatric Abdominal Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NOR001
Record Dates: First submitted 2025-12-02; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Pain Management After Surgery
Keywords: pediatric; TAP-block; postoperative pain management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAP-block (Experimental): Subjects in the TAP-block arm will recieve an open TAP-block at the end of the procedure vbefore wound closure
  Interventions: Procedure: TAP-block
- Wound infiltration (Active Comparator): Subjects in the wound infiltration group will recieve contionious administration of local anastethic via a wound catheter placed subcutaneousley during wound closure.
  Interventions: Procedure: Wound catheter

INTERVENTIONS:
Procedure: TAP-block — Open TAP(transverse abdominal plane)-block placed by the surgeon using open technique at end of surgery before wound closure
  Arms: TAP-block
Procedure: Wound catheter — A catheter placed subcutainiousley for the continuous administration of local anestethic in the wound for up to 3 days post-op
  Arms: Wound infiltration

SUMMARY:
The goal of this trial is to evaluate an open TAP-block vs continuous administration of local anestetic via a wound catheter for postoperative pain management in patients 1-15 years of age undergoing open abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 1-15 years
* Scheduled for elective or acute open adominal surgical procedure

Exclusion Criteria:

* chronic abdominal pain
* known allergy to local analgetic
* Stage 4 renal failure
* psychiatric ailnment

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 88 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative opiates | during the first 24 hours following surgery and total opioids until discarge up to 14 days postoperative
  Amount of postoperative opiates administered

SECONDARY OUTCOMES:
Lenght of stay | Days from surgery through study completeion, an average expected time of7 days
  Duration of hospital stay
Pain assessment | End of surgery until 24 hours post-op
  Pain assesment using validated instruments, FLACC or FPS-R

CONTACTS AND LOCATIONS:
Overall Officials: Oskar Nensén, MD, PhD, Principal Investigator — Uppsala University
Locations (1):
- Akademiska sjukhuset, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: Yes
IPD (anonymized) underlying data in a future publication will be made available on request.